CLINICAL TRIAL: NCT00281515
Title: An Open-label, Multicenter, Randomized Phase II Study to Compare the Effects of Paclitaxel/Carboplatin and Lonafarnib to Those of Paclitaxel/Carboplatin for First-line Treatment of Patients With Epithelial Ovarian Cancer FIGO Stages IIB-IV
Brief Title: Comparison of Paclitaxel/Carboplatin and Lonafarnib to Paclitaxel/Carboplatin for First-line Treatment of Ovarian Cancer
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: AGO Study Group (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Factorial | Masking: None | Purpose: Treatment
Other Study IDs: AGO-OVAR 15
Record Dates: First submitted 2006-01-24; First posted 2006-01-25 (Estimated); Last update posted 2012-06-29 (Estimated); Status verified 2012-06

CONDITIONS: Epithelial Ovarian Cancer
MeSH Terms: conditions — Carcinoma, Ovarian Epithelial | interventions — lonafarnib

ARMS (2):
- Lonafarnib / Paclitaxel /Carboplatin (Experimental)
  Interventions: Drug: Lonafarnib
- Paclitaxel/Carboplatin (Other): Standard Chemotherapy
  Interventions: Drug: Lonafarnib

INTERVENTIONS:
Drug: Lonafarnib — 100mg/twice a day during chemotherapie,in maintenance phase 200 mg twice a day

SUMMARY:
The purpose of this study is to compare the effects of Paclitaxel/Carboplatin and Lonafarnib to those of Paclitaxel/Carboplatin in primary treatment of patients with epithelial ovarian cancer.

DETAILED DESCRIPTION:
Today the standard therapy for patients with advanced ovarian carcinoma is paclitaxel and carboplatin. Lonafarnib is a farnesyl transferase inhibitor (FTI) that is active against a broad spectrum of tumor cell lines in vitro and tumor xenografts in nude mice. Lonafarnib has single-agent antitumor activity as well as enhanced activity in combination with taxanes in a number of tumor cell lines and in vivo models.

ELIGIBILITY:
Inclusion Criteria:

* Previously untreated patients with a histologically confirmed diagnosis of cancer of the ovary, the fallopian tube or extra-ovarian papillary serous tumors FIGO stage IIB-IV, regardless of measurable or non-measurable disease
* Age >= 18 years
* ECOG performance status <= 2
* Life-expectancy of at least 6 months
* Adequate bone marrow, renal and hepatic function:

WBC >= 3.0 x 10^9/l; Neutrophils (ANC) >= 1.5 x 10^9/l; Platelets >= 100 x 10^9/l; Hemoglobin > 6 mmol/l (> 10.0 g/dl); Bilirubin <= 1 x upper limit of normal range; Alkaline phosphatase <= 2.5 x upper limit of normal range; estimated GFR >= 50 ml/min according to Jelliffe or Cockroft-Gault formula

* Patients who have given their signed and written informed consent to participate in the trial after fully understanding the implication and constraints of the protocol
* Patients must be geographically accessible for treatment and follow-up
* Time between definitive surgery and randomization into the study <= 6 weeks

Exclusion Criteria:

* Ovarian tumors of low malignant potential (borderline tumors)
* Non-epithelial ovarian or mixed epithelial/nonepithelial tumors (e.g. Mixed Mullerian tumors)
* Patients who have received previous chemotherapy or radiotherapy
* Prior treatment with FT inhibitors
* Patients with a prior diagnosis of any malignancy not cured by surgery alone less than 5 years before study entry (except in situ carcinoma of the cervix or adequately treated basal cell carcinoma of the skin)
* Complete bowel obstruction or the presence of symptomatic brain metastases
* Concurrent severe medical problems unrelated to malignancy which would significantly limit full compliance with the study or expose the patient to extreme risk or decreased life expectancy
* Patients with a history of seizure disorder or central nervous system disorders; pre-existing motor or sensory neurologic pathology or symptoms > NCI grade 1
* History of congestive heart failure (NYHA Classification > 2, even if medically controlled.
* History of clinical and electrocardiographically documented myocardial infarction within the last 6 months.
* History of atrial or ventricular arrhythmias (>= LOWN II)
* Patients with significant Fridericia QTc (QTcF) prolongation at Baseline (ie. QTcF >= 470 msec)
* Patients with severe active infection
* Patients with a history of severe hypersensitivity reactions to products containing Cremophor EL (cyclosporin or vitamin K) and/or patients with known hypersensitivity to compounds chemically related to Carboplatin and Paclitaxel
* Women with childbearing potential and who are sexually active and unwilling to use a medically acceptable method of contraception (oral contraceptive, diaphragm with spermicide, intrauterine device, condom with spermicide)
* Women who are pregnant or breast feeding
* Administration of other anticancer therapy or simultaneous chemotherapeutic and/or hormonal drugs, or radiotherapy during the study treatment period (except: hormonal replacement therapy and/or steroid antiemetics)
* Patients who are participating in any other clinical study
* Dementia or significantly altered mental status that would prohibit the understanding and giving of informed consent

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 105 (Actual)
Dates: Start 2006-01; Primary Completion 2011-12 (Actual); Study Completion 2011-12 (Actual)

PRIMARY OUTCOMES:
Progression-free survival | every 3 months until PD

SECONDARY OUTCOMES:
Objective tumor response rate (CR/PR (RECIST)) | During whole trial
Duration of response | Until Progression of disease
Overall survival | Until date of death
safety based on nature, frequency and severity of adverse events | During treatment phase until resolution
Predose lonafarnib concentrations | During treatment
PD activity | Assessment

CONTACTS AND LOCATIONS:
Overall Officials: Werner Meier, Prof. Dr., Principal Investigator — Ev. Krankenhaus, Düsseldorf, Germany
Locations (23):
- Germany (23):
  - Charité - Universitätsmedizin Berlin, Campus Virchow-Klinikum, Klinik für Frauenheilkunde, Berlin
  - Klinikum Bremen Mitte, Frauenklinik, Bremen
  - Carl-Gustav-Carus der TU Dresden, Universitäts-Frauenklinik, Dresden
  - Ev. Krankenhaus, Frauenklinik, Düsseldorf
  - Klinik für Frauenheilkunde der Univ. Erlangen, Erlangen
  - Universitätsfrauenklinik, Essen
  - Klinikum der Johann Wolfgang Goethe Universität, Klinik für Frauenheilkunde u. Geburtshilfe, Frankfurt
  - Universitätsklinikum Freiburg, Frauenklinik, Freiburg im Breisgau
  - Kreiskrankenhaus, Frauenklinik, Gifhorn
  - Klinik u. Poliklinik für Gynäkologie und Geburtshilfe, Greifswald
  - Medizinische Hochschule, Hanover
  - St. Vincentius-Krankenhäuser, Karlsruhe
  - Universitätsklinikum Schleswig-Holstein, Campus Kiel, Klinik für Gynäkologie und Geburtshilfe, Kiel
  - Klinik der Otto-von-Guericke Universität, Frauenklinik, Magdeburg
  - Johannes-Gutenberg-Universität, Universitäts-Frauenklinik, Mainz
  - Klinikum der Philipps-Universität Marburg, Klinik für Gynäkologie, Gynäkologische Endokrinologie, Marburg
  - Klinikum Großhadern, Frauenklinik, München
  - Klinikum rechts der Isar der TU München, München
  - Elblandkliniken, Frauenklinik, Radebeul
  - Klinikum Südstadt, Rostock
  - Universitäts-Frauenklinik, Tübingen
  - Universitätsfrauenklinik, Ulm
  - Dr. Horst Schmidt Klinik, Gynäkologie u. Gynäkologische Onkologie, Wiesbaden

REFERENCES:
- [Result] Meier W, du Bois A, Rau J, Gropp-Meier M, Baumann K, Huober J, Wollschlaeger K, Kreienberg R, Canzler U, Schmalfeldt B, Wimberger P, Richter B, Schroder W, Belau A, Stahle A, Burges A, Sehouli J. Randomized phase II trial of carboplatin and paclitaxel with or without lonafarnib in first-line treatment of epithelial ovarian cancer stage IIB-IV. Gynecol Oncol. 2012 Aug;126(2):236-40. doi: 10.1016/j.ygyno.2012.04.050. Epub 2012 May 4. PMID 22564713